CLINICAL TRIAL: NCT02989935
Title: RELVAR Effects on Parasternal Muscle Activity, Diaphragm, and Ventilation in Severe COPD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Paul Easton, Assoc.Prof. University of Calgary, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REB16-0147
Record Dates: First submitted 2016-12-01; First posted 2016-12-12 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Copd
Keywords: respiratory muscle; bronchodilator
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ventilation

STUDY DESIGN:
Intervention Model Description: Study of RELVAR drug effect on respiratory physiology variables including breathing pattern, and EMG.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluticasone vilanterol bronchodilator (Experimental): Inhalation of fluticasone furoate/vilanterol trifenatate, 100 mcg/25 mcg combination, bronchodilator,using standard dry powder inhaler.
  Interventions include ventilation, parasternal EMG, and phrenic magnetic stimulation.
  Interventions: Procedure: Ventilation; Procedure: Parasternal EMG; Procedure: Phrenic magnetic stimulation

INTERVENTIONS:
Procedure: Ventilation — Measurements of ventilation with subjects seated, and breathing across a pneumotachygraph and pressure transducer to measure inspiratory airflow, during both resting and CO2 stimulated breathing.
Procedure: Parasternal EMG — Recordings of electrical activity (EMG) from the parasternal intercostal muscle in the second intercostal space on the upper anterior chest wall adjacent to the sternum.
Procedure: Phrenic magnetic stimulation — Bilateral maximal magnetic stimulation (Magstim) of the phrenic nerves.

SUMMARY:
This study examines the effect of the ultra long acting beta agonist/corticosteroid bronchodilator combination fluticasone furoate/vilanterol trifenatate, on respiratory muscles and ventilation in adults with severe bronchitis or emphysema (COPD).

DETAILED DESCRIPTION:
In adults with severe, minimally reversible bronchitis or emphysema (COPD), there is progressive hyperinflation of the lungs with associated flattening and inefficiency of the major respiratory muscle, the diaphragm. These changes limit physical activity and exercise, and provoke shortness of breath - dyspnea.

These debilitating symptoms are often significantly lessened with ultra long acting combination bronchodilators, even in adults where the bronchodilator does not produce any measurable improvement in either airflow or lung hyperinflation.

This symptomatic improvement in adults with severe, minimally reversible COPD may occur because of a direct benefit of the bronchodilator on respiratory muscles and ventilation.

This study examines the effect of the ultra long acting bronchodilator fluticasone furoate/vilanterol trifenatate upon the upper anterior chest wall respiratory muscles (parasternals), the diaphragm, and breathing pattern.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory, stable severe COPD (GOLD Class III-IV)
* on long acting bronchodilator therapy
* compliant with use of prescribed medications
* fit for minor surgical procedure including intravenous sedation

Exclusion Criteria:

* hypersensitivity to milk proteins
* hypersensitive to fluticasone furoate/vilanterol formulation
* angina or substantial cardiovascular risk
* exacerbation of COPD within the preceding 2 months
* significant non-respiratory system disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Minute ventilation change | 2 hours after fluticasone furoate/vilanterol bronchodilator inhalation.
  Minute ventilation will be averaged and compared, before and then 2 hours after the bronchodilator inhalation.
Parasternal EMG change | 2 hours after fluticasone furoate/vilanterol bronchodilator inhalation.
  Change in moving averaged, EMG continuously recorded from the parasternal intercostal muscle.
Pressure change with phrenic stimulation | 2 hours after fluticasone furoate/vilanterol bronchodilator inhalation.
  Change in recorded mouth pressure during magnetic stimulation of the phrenic nerves.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Easton, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participant physiologic results and measurements publicly presented.
Supporting Information: Study Protocol
Time Frame: During 2020 as final results are available.
Access Criteria: By researcher contact or inquiry

REFERENCES:
- [Background] Easton PA, Hawes HG, Doig CJ, Johnson MW, Yokoba M, Wilde ER. Parasternal muscle activity decreases in severe COPD with salmeterol-fluticasone propionate. Chest. 2010 Mar;137(3):558-65. doi: 10.1378/chest.09-0197. Epub 2009 Oct 9. PMID 19820074